CLINICAL TRIAL: NCT06886711
Title: A Study on the Safety and Efectiveness of Bifidobacterium Bifidum BBi32 in Improving Lntestinal and Lmmune Functions
Brief Title: Research on the Role of Probiotics in Human Intestinal Health
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wecare Probiotics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WK20250306
Record Dates: First submitted 2025-03-08; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Intestinal Microbiota
Keywords: Probiotics; Intestinal Barrier Function
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic group (Active Comparator): Intervention with Bifidobacterium bifidum BBi32 (30 billion CFUday, 3g) was administered daily for 8 weeks.
  Interventions: Dietary Supplement: Probiotic
- Placebo group (Placebo Comparator): Every day to give 3 g maltodextrin intervention for 8 weeks.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — Dietary supplement: Probiotics. The trial period of this study lasts for 2 months(8weeks), during which each participant will have 3 visits (at month 0, month 1, andmonth 2).
  Arms: Probiotic group
Dietary Supplement: Placebo — Dietary supplement: Placebo. The trial period of this study lasts for 2 months(8weeks), during which each participant will have 3 visits (at month 0, month 1, andmonth 2).
  Arms: Placebo group

SUMMARY:
Evaluate the efectiveness and safety of Bifidobacterium bifidum BBi32 as a food supplement compared to a placebo in improving intestinal andimmune functions in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to attend 3 follow-up visits during the intervention period
2. Agree to provide blood, urine, and stool samples twice during the intervention period
3. Good eyesight, able to read and write, and capable of wearing glasses if needed
4. Good hearing and able to fully comprehend all instructions during the intervention

Exclusion Criteria:

1. Presence of digestive diseases, particularly gastrointestinal disorders (e.g., celiac disease, ulcerative colitis, Crohn's disease)
2. History of serious neurological conditions (e.g., epilepsy, stroke, severe head trauma, meningitis within the last 10 years, brain surgery, brain tumor, or prolonged coma-not including general anesthesia)
3. History of or currently receiving treatment for mental health disorders such as alcohol/drug/substance abuse, schizophrenia, psychosis, or bipolar disorder
4. Currently taking medication for depression or low mood
5. Presence of internal organ failure (e.g., heart, liver, or kidney failure)
6. History of radiation therapy or chemotherapy treatments
7. Underwent general anesthesia within the past three years or are scheduled for general anesthesia within the next 3 months during the trial period
8. History of hepatitis (B or C), HIV, or syphilis

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-03-10 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in Fecal Microbiota Composition Before and After Intervention | Baseline (Week 0) and post-intervention (Week 8)
  Fecal microbiota composition will be analyzed using 16S rRNA gene sequencing to assess taxonomic and relative abundance changes.

CONTACTS AND LOCATIONS:
Locations (1):
- Henan University of Technology, Zhengzhou, Henan, China